CLINICAL TRIAL: NCT06347250
Title: A Nerve Block Therapy for Bulbar Palsy Pharyngeal Dysphagia: A Randomized Controlled Study
Brief Title: A Nerve Block Therapy for Bulbar Palsy Pharyngeal Dysphagia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Babujinaya Cela (Other Government)
Responsible Party: Sponsor-Investigator, Babujinaya Cela, Director, Buraidah Central Hospital
Organization: Buraidah Central Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SGB-Bulbar Palsy
Record Dates: First submitted 2024-03-22; First posted 2024-04-04 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-03

CONDITIONS: Bulbar Palsy
MeSH Terms: conditions — Bulbar Palsy, Progressive | interventions — Nerve Block; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nerve block (Experimental): The patients were given Nerve block and routine therapy for 10 days.
  Interventions: Procedure: Nerve Block; Drug: Lidocaine Hydrochloride; Behavioral: routine therapy
- placebo (Placebo Comparator): The patients were given placebo block and routine therapy for 10 days.
  Interventions: Behavioral: routine therapy; Procedure: placebo block

INTERVENTIONS:
Procedure: Nerve Block — The percutaneous approach via the paratracheal route was used for Stellate ganglion block. The operator stood on the side of the block, instructed the patient to lie supine with a thin pillow placed below the shoulders, and tilted the head 45° towards the blocked side, fully exposing the neck. Then, routine disinfection of the neck skin was performed. The puncture site was located 2.5 cm above the sternoclavicular joint and 1.5 cm lateral to the midline of the neck.
  Arms: Nerve block
Drug: Lidocaine Hydrochloride — the patients were provided with Stellate ganglion block, using 1.5ml of 2% Lidocaine hydrochloride (1ml: 0.5mg) and 500ug of Vitamin B12 (1ml: 0.5g).
  Arms: Nerve block
Behavioral: routine therapy — All the participants are provided with the comprehensive rehabilitation (routine rehabilitation and swallowing function training). The routine rehabilitation included intervention for risk factors (blood pressure, blood lipids, blood glucose, smoking and alcohol restriction, exercise, etc.).
  Regrading swallowing function training, both groups are given swallowing function training, including 1) exercises of closure of the vocal folds, pharyngeal, and laryngeal muscles exercises, and respiratory muscle strength training, for 15 min each time and twice per day. 2) isotonic／isometric swallowing exercises, supraglottic swallowing exercises, for 20 min each time and twice per day. 3) effortful swallowing exercises, and cough reflex training, for 10 min each time and twice per day.
Procedure: placebo block — the patients were provided with normal saline. The percutaneous approach via the paratracheal route was used for Stellate ganglion block. The operator stood on the side of the block, instructed the patient to lie supine with a thin pillow placed below the shoulders, and tilted the head 45° towards the blocked side, fully exposing the neck. Then, routine disinfection of the neck skin was performed. The puncture site was located 2.5 cm above the sternoclavicular joint and 1.5 cm lateral to the midline of the neck.
  Arms: placebo

SUMMARY:
This was a multicenter randomized controlled study. 66 post-stroke patients with pharyngeal dysphagia were randomly allocated to the observation group or the control group. Both groups were provided with comprehensive rehabilitation including routine rehabilitation and swallowing function training. Besides, the observation group additionally underwent the stellate ganglion block (SGB). At admission and after 20-day treatment,Yale Pharyngeal Residue Severity Rating Scale, video fluoroscopic swallowing study (VFSS), Functional Oral Intake Scale, and Rosenbek penetration-aspiration scale (PAS) were used to assess swallowing function.

DETAILED DESCRIPTION:
Dysphagia is a frequent and potentially serious complication of stroke. However, there is no effective measure for the treatment of pharyngeal dysphagia in stroke patients. This study aims to explore the efficacy of stellate ganglion block in post-stroke pharyngeal dysphagic patients who received comprehensive rehabilitation. This was a multicenter randomized controlled study. 66 post-stroke patients with pharyngeal dysphagia were randomly allocated to the observation group or the control group. Both groups were provided with comprehensive rehabilitation including routine rehabilitation and swallowing function training. Besides, the observation group additionally underwent the stellate ganglion block (SGB). At admission and after 20-day treatment,Yale Pharyngeal Residue Severity Rating Scale, video fluoroscopic swallowing study (VFSS), Functional Oral Intake Scale, and Rosenbek penetration-aspiration scale (PAS) were used to assess swallowing function.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with ischemic stroke according to the diagnostic criteria, with the stroke occurring in the medulla oblongata and diagnosed as bulbar palsy.
* Upper Esophageal Sphincter did not open or opened ineffectively, with food residue or aspiration, revealed by Videofluoroscopic Swallow Study.
* Age >18 years.
* First-time stroke.
* Steady vital signs,
* Transferred or admitted to the Department of Rehabilitation Medicine within 15d after onset.

Exclusion Criteria:

* Allergy to Lidocaine injection or vitamin B12 injection;
* Severe cognitive impairment;
* Coagulation disorders;
* Severe dysfunction of organs including heart, lungs, kidney, liver, etc.;
* Complicated with other neurological diseases;
* Dysphagia caused by other diseases or reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-05-02 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
The Functional Oral Intake Scale | day 1 and day 10
  The Functional Oral Intake Scale (FOIS) is a tool used to assess the level of independence in oral intake for individuals with swallowing difficulties. The scale ranges from Level 1 to Level 7, with higher Levels indicating better swallowing function.

SECONDARY OUTCOMES:
Yale Pharyngeal Residue Severity Rating Scale | day 1 and day 10
  The Yale Pharyngeal Residue Severity Rating Scale (Yale) was used to assess the severity of pharyngeal residue in patients. While PAS primarily evaluated whether food or liquid entered the airway, Yale focused on the condition of pharyngeal residue. The scale includes the four levels from 0 to 3, with lower levels indicating less severe pharyngeal residue.
penetration-aspiration scale | day 1 and day 10
  this assessment evaluated the patient's swallowing of contrast medium and whether there was retention, penetration, and aspiration. It included multiple items, each with the corresponding criteria, Specifically, whether the swallowed material entered the airway, passed through or contacted the vocal cords, and whether the patient exhibited the corresponding ability to clear. There were 8 levels in the results, with higher levels indicating more severe aspiration.
Video fluoroscopic swallowing study | day 1 and day 10
  The patient was required to take a sitting position with the head naturally upright. Under the guidance of the examiner, the patient first swallowed 5ml of iohexol solution (50ml:17.5g in iodine terms). If the patient exhibited aspiration, the test would stop. If not, the patient was instructed to swallow 10ml of iohexol solution mixed with breadcrumbs, and the patient's swallowing condition was observed with immediate measures ready to take for safety. Specially, the esophageal phase was not included in the study, because it was commonly regarded as an independent phase. The swallowing were divided into 3 phases in this assessment: Oral phase, Pharyngeal phase, and Aspiration, with maximum 3,3,4 points were given to each phase. The total score was calculated as the final result. The final score was positively correlated with the swallowing function.
The Swallowing Quality of Life Questionnaire | day 1 and day 10
  The Swallowing Quality of Life Questionnaire (SWAL-QOL) is a tool designed to assess how swallowing difficulties impact an individual's quality of life. The questionnaire covers various aspects such as eating, speech, and social interaction to understand the challenges and effects of swallowing disorders on daily life.
  SWAL-QOL scores can range from 0 to 100, with higher scores indicating a better quality of life related to swallowing function. Therefore, a higher SWAL-QOL score reflects less negative impact of swallowing difficulties on an individual's overall quality of life, highlighting better adaptation to and management of swallowing issues.

CONTACTS AND LOCATIONS:
Overall Officials: Nieto Luis, Master, Study Director — Site Coordinator of United Medical Group
Locations (1):
- ZhenD No.1 Hos., Zhenzhou, China